CLINICAL TRIAL: NCT00905697
Title: Analysis of Patient Reported Outcomes in Living Donor Lung Transplantation
Brief Title: Patient Reported Outcomes in Living Donor Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Toru Oga, Department of Respiratory Care and Sleep Control Medicine, Kyoto University, Graduate School of Medicine
Other Study IDs: E561kyoto
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lung Transplantation
Keywords: Living donor lung transplantation; Health-related quality of life; Prognosis; Patient reported outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Living donor lung transplantation: Living lung transplantation donors
  Interventions: Procedure: Living donor lung transplantation

INTERVENTIONS:
Procedure: Living donor lung transplantation — Living donor lung transplantation

SUMMARY:
The purpose of the present study is to investigate how the health of donors in living donor lung transplantation will change after transplant operations.

DETAILED DESCRIPTION:
In Japan, living donor lung transplantation has been established as an alternative therapy for brain-dead lung transplantation, as the number of organs for transplantation is absolutely short. However, how patient reported measurements including health status, dyspnea, psychological status and sleep would change after lung transplantation has not been well evaluated. Therefore, in the present study, we aim (1) to compare them before and after transplant operations and (2) to analyze how they will change for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* New donors for living donor lung transplantation

Exclusion Criteria:

* Inability to obtain informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kyoto University Hospital Clinic for Lung Transplantation
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in health status | At entry and every year for 5 years

SECONDARY OUTCOMES:
Change in dyspnea | At entry and every year for 5 years
Change in psychological status | At entry and every year for 5 years
Change in sleep quality | At entry and every year for 5 years
Prognosis | At entry and every year for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Date, MD, PhD, Study Chair — Graduate School of Medicine, Kyoto University
Locations (1):
- Graduate School of Medicine, Kyoto University, Kyoto, Japan